CLINICAL TRIAL: NCT07403812
Title: Assessing the Performance of "DCog Short", an iPad-Based Tool for Neurotoxicity Evaluation in CAR-T Cell Therapy Patients: A Pilot Study
Brief Title: Assessing DCog Short for Neurotoxicity in CAR-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jon Arnason, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-610
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Neurotoxicity; Neurotoxicity Syndromes; Hematologic Malignancy; Immune Effector Cell Associated Neurotoxicity Syndrome
Keywords: Neurotoxicity; Neurotoxicity Syndrome; Hematologic Malignancy; Immune Effector Cell Associated Neurotoxicity Syndrome
MeSH Terms: conditions — Neurotoxicity Syndromes; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CAR-T Cell Therapy Patients (Experimental): 40 enrolled participants will complete:
  * Baseline visit
  * Daily study visits during hospitalization, then via phone: 2x weekly on days 14 - 21, then weekly on days 21 - 30
  * 90 Day follow up visit
  Interventions: Behavioral: DCog Short

INTERVENTIONS:
Behavioral: DCog Short — An iPad-based cognitive assessment instrument to evaluate neurotoxicity and consisting of a series of tests that measure various aspects of cognitive function. After hospital discharge, participants will be provided with iPads which will be returned at the 90 day follow up visit.

SUMMARY:
The aim of this study is to determine the effectiveness of DCog Short, a self-reporting, iPad-based application tool, in assessing neurotoxicity in participants undergoing CAR-T cell therapy.

DETAILED DESCRIPTION:
The goal of this pilot study is to determine the effectiveness of DCog Short, a self-reporting, iPad-based application tool, in assessing neurotoxicity in participants undergoing CAR-T cell therapy. This is the first time investigators are examining this tool.

The U.S. Food and Drug Administration (FDA) has not approved DCOG Short as a mobile application tool to evaluate neurotoxicity for hematologic malignancies.

The research study procedures include screening for eligibility, questionnaires, and cognitive assessments.

It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* participants treated with CART-Cell therapy as described above and therefore at risk for treatment associated neurotoxicity.
* Visual acuity of 20/100 or better.

Exclusion Criteria:

* patients < 18 years old
* pregnant women
* prisoners
* adults unable to consent,
* participants unwilling to use iPad-based tools. Severe motor deficits that can prevent patients from using an iPad

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of DCog Short for Early Detection of Neurotoxicity | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  Neurotoxicity is defined as any decrease from 10 on the Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) 10-point scale, where 10 indicates no impairment. The DCog Short assessment will be compared with the standard clinical ICANS evaluation to determine its ability to detect neurotoxicity on or before the onset of clinically confirmed ICANS. Sensitivity is defined as the proportion of patients with clinically confirmed ICANS for whom DCog Short indicates neurotoxicity on or before ICANS onset. DCog Short will be considered effective if sensitivity is ≥75% and non-promising if sensitivity is <50%.
Specificity of DCog Short for Early Detection of Neurotoxicity | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  Neurotoxicity is defined as any decrease from 10 on the Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) 10-point scale, where 10 indicates no impairment. The DCog Short assessment will be compared with the standard clinical ICANS evaluation to determine its ability to correctly identify patients who do not develop neurotoxicity. Specificity is defined as the proportion of patients who do not develop clinically confirmed ICANS and are not indicated by DCog Short. DCog Short will be considered effective if specificity is ≥75% and non-promising if specificity is <50%.
Positive Predictive Value (PPV) of DCog Short for Early Detection of Neurotoxicity | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  Neurotoxicity is defined as any decrease from 10 on the Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) 10-point scale, where 10 indicates no impairment. The DCog Short assessment will be compared with the standard clinical ICANS evaluation to determine its ability to correctly identify patients who do not develop neurotoxicity. Positive predictive value is defined as the proportion of patients indicated by DCog Short who subsequently develop Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) based on standard clinical assessment.
Negative Predictive Value (NPV) of DCog Short for Early Detection of Neurotoxicity | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  Neurotoxicity is defined as any decrease from 10 on the Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) 10-point scale, where 10 indicates no impairment. The DCog Short assessment will be compared with the standard clinical ICANS evaluation to determine its ability to correctly identify patients who do not develop neurotoxicity. Negative predictive value is defined as the proportion of patients not indicated by DCog Short who do not develop Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) based on standard clinical assessment.
Raw Accuracy of DCog Short for Early Detection of Neurotoxicity | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  Neurotoxicity is defined as any decrease from 10 on the Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) 10-point scale, where 10 indicates no impairment. The DCog Short assessment will be compared with the standard clinical ICANS evaluation to determine its ability to correctly identify patients who do not develop neurotoxicity. Raw accuracy is defined as the proportion of patients correctly classified by DCog Short, including both patients who develop Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) and those who do not, based on standard clinical assessment.

SECONDARY OUTCOMES:
Immune Effector Cell-Associated Encephalopathy (CARTOX-10) Score Change from Baseline | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  For ICANS detection and monitoring, the Immune Effector Cell-Associated Encephalopathy (ICE) score, also called CARTOX-10, will be used. The total score ranges from 0 to 10, with higher scores indicating normal cognitive function. Detailed scoring instructions and grading criteria are provided in Appendix A of the protocol.
Differences in Neurotoxicity Development and Detection Across CAR T-Cell Therapy Types | Until 30 days post CAR T-cell infusion, with frequency as described in the protocol schedule section 10.0.
  Neurotoxicity will be monitored using DCog Short and CARTOX-10 assessments throughout the study period. Immune Effector Cell-Associated Encephalopathy (ICE) score, e ranges from 0 to 10, with higher scores indicating normal cognitive function. Detailed scoring instructions and grading criteria are provided in Appendix A of the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Arnason, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu